CLINICAL TRIAL: NCT00827866
Title: Efficacy of Tobacco Quitline for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: XPD07-140 Quit-Line; R01CA127964 (NIH)
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2014-11

CONDITIONS: Smoking Cessation
Keywords: Tobacco quitline; Childhood cancer survivors; Adult-onset cancer survivors
MeSH Terms: conditions — Smoking Cessation | interventions — DMAC2L protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Counselor-Initiated Tobacco Quit Line Group QL where the counselor contacts the client with a standardized intervention protocol)
  Interventions: Other: Counselor-Initiated Tobacco Quit Line
- 2 (Other): Self-Paced Tobacco Quit Line Group which leaves the calling up to participants
  Interventions: Other: Self-Paced Tobacco Quit Line

INTERVENTIONS:
Other: Counselor-Initiated Tobacco Quit Line — The proposed active intervention will be a the Counselor-Initiated QL which includes provision of 8 weeks of nicotine replacement therapy (NRT) and six scheduled telephone sessions of a behavioral intervention.
  Other Names: Other: Arm 1
  Arms: 1
Other: Self-Paced Tobacco Quit Line — The comparison condition will be the Self-Paced QL with provision of 2 weeks of NRT and encouraged obtainment of additional NRT. If participants in the Self-Paced condition make all six calls, they will receive the same behavioral intervention as in the Counselor-Initiated condition.
  Other Names: Arm 2
  Arms: 2

SUMMARY:
The proposed study is a two-armed randomized controlled clinical trial examining the long-term (one-year) efficacy of telephone intervention conditions for smoking cessation in a high risk medical population; namely, cancer survivors: Proactive telephone recruitment through the Childhood Cancer Survivors Survey (CCSS) St. Jude Life Study, After Completion of Therapy (ACT) Clinic and face to face recruitment at the local West Clinics will serve as the primary methods of recruitment.

The specific aims of the study :

(1) To recruit nationally a cohort of approximately 1242 smokers who are cancer survivors(621 childhood cancer survivors and 621 adult cancer survivors); 2) To determine the long-term (one year) efficacy of the intervention condition for participants randomly assigned to the Counselor-initiated versus a Self-paced QL; and (3) to find out whether treatment outcomes vary as a function of survivors' age of cancer diagnosis (survivors who diagnosed while adults vs. childhood cancer survivors who diagnosed before the age of 21).

DETAILED DESCRIPTION:
In this study participants (n=1242) will be randomly assigned to a Counselor-Initiated Tobacco Quit Line (QL;) in which the counselor contacts the client with the standardized intervention protocol, or a Self-Paced Tobacco QL (which leaves the calling up to participants).The proposed active intervention will be a the Counselor-Initiated QL which includes 8 weeks of nicotine replacement therapy (NRT) and six scheduled telephone sessions of a behavioral intervention. The comparison condition will be the Self-Paced QL with provision of 2 weeks of NRT and encouraged obtainment of additional NRT. If participants in the Self-Paced condition make all six calls, they will receive the same behavioral intervention as in the Counselor-Initiated condition.

ELIGIBILITY:
Inclusion Criteria:

* Participants smokes cigarettes
* Participants is a cancer survivor
* Participant must be at least 18 years of age.
* Childhood cancer survivors must be at least one year out active cancer treatment.
* Participant understands consent procedures.
* Participant speaks English.
* Participant must have access to a telephone for participation

Exclusion Criteria:

* Inability to understand consent procedures
* Participants with a known contraindication or sensitivity to nicotine replacement therapy may participate in this study; however they will not receive nicotine replacement therapy (NRT) as part of their smoking cessation program.
* Since our participants are childhood cancer survivors and they can be medically fragile and we are interested in providing all eligible participants with NRT to enhance their ability to quit smoking, we added a cautionary conditions list to the recruitment screening form. Those with severe arrhythmias, myocardial infarction, unstable angina, cerebrovascular incident, blood vessel disease, phaeochromocytoma, diabetes, hyperthyroidism, abnormal kidney or liver function, or history of gastritis or peptic ulcers, or who smoke less than 5 cigarettes per day will not receive NRT.
* Patients with questionable NRT eligibility will be discussed/reviewed on a case by case basis with the Staff Family Physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 946 (Actual)
Dates: Start 2008-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Self-reported prolonged abstinence and cotinine-validated point-prevalence abstinence at 1 year follow-up | 1 year

SECONDARY OUTCOMES:
Account for dose of treatment (NRT use plus number of QL contact) vs. success(quit for one year response) independent of treatment assignment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Klesges, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Derived] Klesges RC, Krukowski RA, Klosky JL, Liu W, Srivastava DK, Boyett JM, Lanctot JQ, Hudson MM, Folsom C, Lando H, Robison LL. Efficacy of a tobacco quitline among adult cancer survivors. Prev Med. 2015 Apr;73:22-7. doi: 10.1016/j.ypmed.2014.12.019. Epub 2015 Jan 5. PMID 25572620
- See also: St. Jude Children's Research Hospital — http://www.stjude.org